CLINICAL TRIAL: NCT04065217
Title: Diode Laser 980-nm in Hemangioma Treatment
Brief Title: The Effectiveness of Diode Laser 980-nm in Iraqi Face Hemangioma: a Randomized Within Patients Trial
Acronym: NTDL980
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noor Taha Ismaeel (Other)
Responsible Party: Sponsor-Investigator, Noor Taha Ismaeel, Assistant Lecturer, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1477
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hemangioma
Keywords: Hemangioma; Randomized within patient; Diode laser; Histogram
MeSH Terms: conditions — Hemangioma | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: uni-center, government clinic, randomized within patient trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iraqi patients with face hemangioma (Other): Diode laser 980-nm in the diseased group only while we no need the comparator group because we compared between lesion before and after. The administration of laser is scheduled to start treatment. Patients will take laser therapy as a 12 session at two week-interval. In case of intolerance, session number reduction by 10, 8, 6, 4 allowed. Adherence to treatment will be assessed at each interval for undesired side effects or complications. The intervention should continue also after complete session, or during temporary interval withdrawal due to reached maximal cumulative response or side effects from laser therapy.
  Interventions: Procedure: Diode laser 980-nm

INTERVENTIONS:
Procedure: Diode laser 980-nm — Before starting the laser session, cosmetics or makeup were removed and the skin was cleaned. The area was anesthetized by the application of as EMLA lotion (lidocaine 2.5% + prilocaine 2.5%) [ONLY MEDICAL; CAT No. R331/72394/P001] 20 minutes before the session. During the procedure, the laser probe was held perpendicular to the lesion and a guide beam was used to direct the application. The patient wore protective eye goggles [CE; DIR 8001100L4]. After the session, cool air was applied to the whole region. Each patient received a maximum of six sessions, delivered at two-week intervals. Patients reported itchiness and erythema during the session.

SUMMARY:
In an academic, government clinic, uni-center, randomized within patients trial study of the effects of 980-nm diode laser treatment included 15 cases of facial hemangiomas in patients with a history of discomfort due to lesions that were not suitable for removal using traditional methods. The study was carried out at the University of Baghdad/Institute of Laser for Postgraduate Studies/Laser Medicine Research Clinics from 15 October 2018 to 15 April 2019. Primary end-point is improvement of conditions at 6 months. Secondary end-points are quality of life, disappear lesions and safety administration of diode laser. Each patient received 12 sessions at two-week intervals. Lesions were photographed before and after laser treatment and digital image histograms were generated as a graphical representation of the tonal distribution.

Following treatment, the lesions were less elevated, smoother in texture, and the color changed from dark red to light pink.

There is a need to improve the treatment of face hemangiomas. Results from this randomized within patient trial will serve as preliminary evidence of the future role of diode laser in hemangioma treatment and a basis for design and power estimations of future studies. Based on the skin texture, color and elevation of the hemangioma as well as patient satisfaction, this type of laser is a safe and effective modality for the treatment of facial hemangioma in Iraqi patients.

ELIGIBILITY:
Inclusion Criteria:

1. Comfortable.
2. Superficial lesion.

Exclusion Criteria:

1. Advanced case.
2. Deep lesion.
3. Uncomfortable.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Area of Hemangioma lesions | 4th week
  Measured area of lesions by tape measure by centimeters
Color of lesion | 4 weeks
  By inspection color of lesion change from dark red to bright red or disappear
Shape of lesion | 4 weeks
  Clinical exam by inspection, we look to ugly shape of lesion, may be change for better or disappear

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Laser for Postgraduate Studies, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Data availability
Supporting Information: Study Protocol, SAP, CSR
Time Frame: one year
Access Criteria: Open
URL: http://doi.org/10.5281/zenodo.3338657